CLINICAL TRIAL: NCT00682058
Title: Body Composition & REE Responses to Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dympna Gallagher, Associate Professor of Nutritional Medicine, Columbia University
Other Study IDs: AAAO1655; R01DK072507 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Weight Loss; Weight Change
Keywords: body composition; weight loss; fat; fat distribution; fat free mass; organ; resting energy expenditure
MeSH Terms: conditions — Weight Loss; Body Weight Changes; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LABS patients: Bariatric surgery patients with 35>BMI kg/m2<60 prior to surgery will undergo follow-up post-bariatric surgery.
  Interventions: Other: Follow-up post-bariatric surgery

INTERVENTIONS:
Other: Follow-up post-bariatric surgery — Follow-up of those subjects who had bariatric surgery (as part of the parent LABS trial) immediately following the collection of baseline measures (body composition) in this study. Follow-up body composition measures will be acquired at 60 months and 84 months post-baseline measures (post-surgery).
  Other Names: Observational at this time with no intervention

SUMMARY:
The aim of this study is to measure important components of weight change in patients who underwent bariatric surgery on measures of fat mass and its distribution and fat-free mass (FFM) (bone mineral density, skeletal muscle, and specific organs) at 60 months (T60) and 84 months (T84) post-surgery, and to compare compartment sizes with stable weight controls.

DETAILED DESCRIPTION:
Consenting, eligible patients previously enrolled in the ancillary study, "Longitudinal Assessment of Bariatric Surgery" (LABS), from Weill Cornell and the University of Pittsburgh will undergo the following measures: total body water by deuterium dilution (fat and fat-free mass (FFM)), extracellular water by sodium bromide tracer, body density by the BodPod, whole-body magnetic resonance imaging (MRI) (adipose tissue and its distribution; skeletal muscle mass; mass of liver, kidneys, heart, and brain), dual energy-X-ray absorptiometry (femur bone mineral density (BMD), total body fat, fat-free mass, and bone mineral content), and resting energy expenditure (REE). MRI will describe body composition changes at the tissue/organ level and adipose tissue distribution allowing us to address questions of biological and clinical importance including the body composition changes' influences on REE. The specific aims are to: 1) measure important components of weight change in patients who underwent bariatric surgery on measures of fat mass and its distribution and FFM (including bone mineral density, skeletal muscle, and specific organs) at T60 and T84 months following surgery, and also to compare compartment sizes with those seen in stable weight controls; 2) measure the amount of change in REE at T60 and T84 compared to T0, following weight loss induced by bariatric surgery and to determine its relation to changes in body composition compartments, and its duration over the follow-up period. Secondary research questions relate to changes in cardiac structure and function, physical activity associations with skeletal muscle changes, and adipose tissue depot changes as predictors of cardiometabolic parameters (glucose metabolism and serum lipid composition). Subjects will be women and men (n=100) equally distributed between the New York and Pittsburgh sites.

ELIGIBILITY:
* Had to have been enrolled in the ancillary study prior to having bariatric surgery
* Are able to come to the laboratory for testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consented and enrolled in the ancillary study, LABS, prior to having bariatric surgery; all came from Weill Cornell and the University of Pittsburgh LABS sites
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2006-10; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Fat and fat-free mass | Approximately 60 months and 84 months post-bariatric surgery

SECONDARY OUTCOMES:
Adipose tissue distribution | Approximately 60 months and 84 months post-bariatric surgery

OTHER OUTCOMES:
Resting energy expenditure | Approximately 60 months and 84 months post-bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: James Delany, PhD, Study Director — University of Pittsburgh
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ashby-Thompson M, Heshka S, Rizkalla B, Zurlo R, Lemos T, Janumala I, Goodpaster B, DeLany J, Courcoulas A, Strain G, Pomp A, Kang P, Lin S, Thornton J, Gallagher D. Validity of dual-energy x-ray absorptiometry for estimation of visceral adipose tissue and visceral adipose tissue change after surgery-induced weight loss in women with severe obesity. Obesity (Silver Spring). 2022 May;30(5):1057-1065. doi: 10.1002/oby.23415. Epub 2022 Apr 6. PMID 35384351